CLINICAL TRIAL: NCT04895423
Title: Evaluation of the Effectiveness and Safety of Immunosuppressive and Biological Therapy of Atopic Dermatitis in Childhood
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04532781
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Atopic Dermatitis
Keywords: Glucocorticoids; Biologic Drugs; Methotrexate; Cyclosporine; dupilumab
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group №1: Methotrexate therapy (Experimental)
  Interventions: Drug: Methotrexate therapy
- Group №2: Mycophenolate mofetil therapy (Experimental)
  Interventions: Drug: Mycophenolate mofetil therapy
- Group №3: Cyclosporine therapy (Experimental)
  Interventions: Drug: Cyclosporine therapy
- Group №4: Dupilumab therapy (Experimental)
  Interventions: Drug: Dupilumab therapy

INTERVENTIONS:
Drug: Methotrexate therapy — Methotrexate subcutaneously 10-15 mg/m2 once every 7 days within 12 months
  Arms: Group №1: Methotrexate therapy
Drug: Mycophenolate mofetil therapy — Mycophenolate mofetil per os 500-700 mg/m2 2 times a day within 12 months
  Arms: Group №2: Mycophenolate mofetil therapy
Drug: Cyclosporine therapy — Cyclosporine per os 3 mg/m2 2 times a day within 12 months
  Arms: Group №3: Cyclosporine therapy
Drug: Dupilumab therapy — Patients weighing <30 kg received an initial dose of 600 mg (2 injections of 300 mg subcutaneously), then 300 mg every 4 weeks. Patients weighing 30 to <60 kg received an initial dose of 400 mg (2 injections of 200 mg subcutaneously), then 200 mg every 2 weeks; Patients weighing 60 kg or more, the initial dose is 600 mg (2 injections of 300 mg subcutaneously), then 300 mg every 2 weeks.
  Arms: Group №4: Dupilumab therapy

SUMMARY:
This comparative study analyzes the efficacy and safety of treatment of children from 6 years of age suffering from moderate to severe atopic dermatitis using an inhibitor of IL4, IL13 and classical immunosuppressants.

DETAILED DESCRIPTION:
This is a prospective study aimed at direct comparative analysis of the efficacy and safety of treatment of children from 6 years of age suffering from moderate and severe atopic dermatitis using a genetically engineered biological drug and classical immunosuppressants.

Based on clinical and anamnestic data, compliance with the inclusion / exclusion criteria, the study included 160 patients from 6 years old, with moderate / severe atopic dermatitis.

The initial indices were assessed: SCORAD- Scoring of Atopic Dermatitis (index for assessing the severity of atopic dermatitis); NRS- numeric rating scale for itch; CDLQI - The Children's Dermatology Life Quality Index; POEM- Patient-Oriented Eczema Measure (personalized assessment of eczema) and laboratory parameters: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, lactate dehydrogenase, gamma-glutamyltransferase, total bilirubin, direct bilirubin, serum albumin, blood urea specific IgE to food and household allergens, indicators of a clinical blood test, indicators of a general analysis of urine, indicators of a biochemical analysis of urine (creatinine, urea).

In the presence of concomitant allergic pathology (bronchial asthma, allergic rhinitis), the CSMS [Combined Symptom and Medication Score] were additionally assessed (Scale for assessing nasal symptoms of rhinitis, taking into account the need for medication); VAS - Visual Analog Scale (visual analog scale); ACT- Asthma Control Test. Subsequently, systemic therapy was prescribed: metorexat (40 people), mycophenolate mofetil (40 people), cyclosporine (40 people) dupilumab (40 people).

ELIGIBILITY:
Inclusion Criteria:

1. Age over 6 years inclusive;
2. Atopic dermatitis diagnosed at least 12 months before the start of the study;
3. Atopic dermatitis of moderate or severe course;
4. Consent to discontinue the use of the following prohibited drugs or any of the following therapies at least 4 weeks before the start of the study and not to use them throughout the study, unless otherwise specified below:

   1. Oral systemic corticosteroids;
   2. Other systemic immunosuppressive drugs;
   3. Phototherapy, including therapeutic phototherapy (psoralen plus ultraviolet A, ultraviolet B), excimer laser, and self-medication using a tanning bed;
5. A signed and dated informed consent received from the patient's parents (guardians), as well as from a patient over 14 years of age, to participate in the study.
6. Ability to attend control visits within the specified time frame

Exclusion Criteria:

1. Use of other genetically engineered biological preparations in therapy;
2. Participation in other clinical trials;
3. The presence of other concomitant skin diseases in the present or in the past, which could affect the assessment of the effect of the study drugs on the course of atopic dermatitis;
4. The presence of herpetic eczema within 12 months before the start of the study;
5. A history of two or more cases of herpetic eczema;
6. The presence in the present of a skin infection for which is required or is being treated with antibiotics for topical use or systemic antibiotics;
7. Therapy with the following drugs:

   1. Other genetically engineered biological preparations less than 5 half-lives before the start of the study.
   2. Any corticosteroid for oral and parenteral administration and administration, which were in therapy for 2 weeks before enrollment in the study, or the possible need for parenteral injection of corticosteroids during the course of the study.
   3. Intra-articular corticosteroid injection within 2 weeks prior to study enrollment; Note: The use of intranasal or inhaled steroids is permitted throughout the study.
8. Extensive or complete disability, significantly limiting personal care or determining the inability to carry it out.
9. Immunodeficiency disease;
10. The presence in the past or present of any serious and / or unstable disease, which, in the opinion of the investigator, may pose an unacceptable risk to the patient in the case of the use of the investigational drug or interfere with the interpretation of the data;
11. History of lymphoproliferative disease; or manifestations or symptoms suggesting the possible presence of lymphoproliferative disease, including lymphadenopathy or splenomegaly; either primary or recurrent malignant disease in active form; or remission after a clinically significant malignant disease lasting less than 5 years;
12. The course of a viral, bacterial, fungal or parasitic infection;
13. Failure or unwillingness of the patient or patient's parent / caregiver / patient legal guardian to comply with the requirements of research participants throughout the study and / or unwillingness to follow research restrictions / procedures, including the use of data loggers.
14. Contraindications to the use of adrenaline.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-11-25 (Estimated); Primary Completion 2023-07-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
SCORAD (Scoring of Atopic Dermatitis) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the SCORAD index
NRS (Numeric rating scale for itch) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the NRS
Adverse events | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  Adverse events monitoring

SECONDARY OUTCOMES:
CDLQI (The Children's Dermatology Life Quality Index) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the CDLQI
POEM (Patient-Oriented Eczema Measure) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the POEM
CSMS (Combined Symptom and Medication Score) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the CSMS
VAS (Visual Analog Scale) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the VAS
ACT (Asthma Control Test) | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change of the ACT
Concentration in the biochemical blood test of total IgE and specific IgE for food and household allergens | screening (baseline), 3, 4, 6 and 12 months from the start of therapy
  change in the Concentration in the biochemical blood test of total IgE, specific IgE-method ImmunoCap to food and household allergens

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided